CLINICAL TRIAL: NCT05319106
Title: Transplantation of Human Umbilical Cord Derived Mesenchymal Stem Cell for Refractory Skin Ulcer Therapy
Brief Title: Phase Ⅱ Clinical Study of Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Venous Leg
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ShiCang Yu (Other)
Responsible Party: Sponsor-Investigator, ShiCang Yu, Director, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zsyx1
Record Dates: First submitted 2022-03-18; First posted 2022-04-08 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Venous Leg Ulcer
Keywords: Venous leg ulcer; human umbilical cord mesenchymal stem cells; wound healing
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stem cell preparation combined with silver ion dressing (Experimental)
  Interventions: Other: stem cell preparation combined with silver ion dressing
- silver ion dressing (Placebo Comparator)
  Interventions: Procedure: silver ion dressing

INTERVENTIONS:
Other: stem cell preparation combined with silver ion dressing — The dosage range of each cm2 ulcer wound is (1～5)×10^6. The dosage of human umbilical cord mesenchymal stem cells for the second treatment is determined according to the severity of the ulcer. Each patient is treated for 2 consecutive times, and the interval between each treatment is 3 days.
  Arms: Stem cell preparation combined with silver ion dressing
Procedure: silver ion dressing — fter wound debridement, a silver ion dressing suitable for the size of the wound was cut and covered on the wound bed. Sterile gauze was covered on the silver ion dressing and fixed with adhesive tape.
  Arms: silver ion dressing

SUMMARY:
This project adopts a prospective clinical trial study to compare and evaluate the efficacy of local transplantation of human umbilical cord mesenchymal stem cells combined with silver ion dressing and simple silver ion dressing in the treatment of venous lower extremity ulcer wounds. To improve the healing rate and quality of life of patients.

DETAILED DESCRIPTION:
Chronic wounds refer to the pathological changes such as cell senescence, imbalance of synthesis and degradation of extracellular matrix, and decreased activity of growth factors caused by different reasons when the wound is prolonged and does not heal after conventional treatment for more than 1 month without healing tendency. Chronic wound can be caused by a variety of diseases, including arterial disease, diabetes, vasculitis, venous disease and skin malignant tumor, chronic venous insufficiency (CVI) is a disease leading to chronic wound, Venous ulcer (VLU) of lower limbs is the advanced manifestation of CVI, and the incidence of this disease ranges from 0.4% to 1.3% in China. 60% of VLU patients' ulcer wounds heal in 3-6 months, 33% in 12 months, and 7% May be permanently unhealed. The probability of recurrence is as high as 70% in patients 3-5 months after wound healing, which not only seriously affects the health and quality of life of patients, but also causes a very heavy social medical burden. At present, the conventional treatment for VLU mainly includes drug therapy, stress therapy, wound treatment and surgical treatment, but the therapeutic effect is not ideal.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 70, no gender limitation;
2. It met the diagnostic criteria of venous ulcer of lower limbs in Clinical Vascular Surgery (5th edition), and the following conditions were met: the ulcer lasted for more than 1 month; The wound area was between 10cm2 and 40cm2. Wound depth: All wounds were deep tissue ulcers below the epidermis.
3. Participate in the clinical study voluntarily, observe the study procedure, and observe the curative effect cooperatively.

Exclusion Criteria:

1. Pregnant or lactation women; Women who have planned to have children recently (within 6 months);
2. Patients with peripheral artery disease with ankle-brachial index (ABI) < 0.8;
3. Patients with active clinical systemic infection;
4. Serious skin wound infection is not under control;
5. low immune function and systemic failure; Severe heart, liver, lung, kidney and other important organ lesions (ALT, AST, Cr & GT; Normal 1.5 times, congestive heart failure ejection fraction < Normal 30%) and severely impaired hematopoietic function;
6. Abnormal coagulation function or current anticoagulant treatment;
7. Systemic autoimmune diseases in the active stage;
8. With systemic organ or hematological malignancy;
9. PERSONS infected with HIV or addicted to drugs, tobacco and alcohol;
10. Have a clear history of mental illness;
11. Participation in clinical studies of any drug within 1 month prior to treatment (or the 5 half-life of the investigational drug, whichever is longer).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Healing time | Epithelialization of the wound completely or 24 weeks after treatment
  The time required for the wound healing rate to reach 100%

SECONDARY OUTCOMES:
Wound shrinkage rate | Epithelialization of the wound completely or 24 weeks after treatment
  Grid method was used to calculate the wound area, with 1 decimal place behind the length unit and 2 decimal places behind the area unit. The wound edges before, during and after treatment were depicted on the transparent mesh film respectively, and the original wound area and the unhealed wound area were calculated.
  Wound shrinkage rate = (initial area of wound - area measured on the day)/original area of wound × 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Army Medical University (Third Military Medical University), Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvarez OM, Markowitz L, Parker R, Wendelken ME. Faster Healing and a Lower Rate of Recurrence of Venous Ulcers Treated With Intermittent Pneumatic Compression: Results of a Randomized Controlled Trial. Eplasty. 2020 Jun 5;20:e6. eCollection 2020. PMID 32636985
- [Result] Nicolaides AN. The Most Severe Stage of Chronic Venous Disease: An Update on the Management of Patients with Venous Leg Ulcers. Adv Ther. 2020 Feb;37(Suppl 1):19-24. doi: 10.1007/s12325-020-01219-y. Epub 2020 Jan 22. PMID 31970660
- [Result] Aleksandrowicz H, Owczarczyk-Saczonek A, Placek W. Venous Leg Ulcers: Advanced Therapies and New Technologies. Biomedicines. 2021 Oct 29;9(11):1569. doi: 10.3390/biomedicines9111569. PMID 34829797
- [Result] Kavala AA, Turkyilmaz S. Autogenously derived regenerative cell therapy for venous leg ulcers. Arch Med Sci Atheroscler Dis. 2018 Dec 15;3:e156-e163. doi: 10.5114/amsad.2018.81000. eCollection 2018. PMID 30775606
- [Result] Zollino I, Campioni D, Sibilla MG, Tessari M, Malagoni AM, Zamboni P. A phase II randomized clinical trial for the treatment of recalcitrant chronic leg ulcers using centrifuged adipose tissue containing progenitor cells. Cytotherapy. 2019 Feb;21(2):200-211. doi: 10.1016/j.jcyt.2018.10.012. Epub 2018 Dec 22. PMID 30583949